CLINICAL TRIAL: NCT03433846
Title: Predictors of Sepsis in Ex-Preterm Infants
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Amy O'Connell, MD, PhD, Boston Children's Hospital
Other Study IDs: IRB-P00023454
Record Dates: First submitted 2018-02-03; First posted 2018-02-15 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Sepsis; Premature Birth
Keywords: Sepsis; Prematurity
MeSH Terms: conditions — Sepsis; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will have up to 0.5 ml of blood collected as a sample within the first 1-2 weeks after the subject is enrolled. After that any discard blood samples which have been obtained as part of clinically requested blood draws will be obtained from the Core Laboratory at the institution.
  If there are no discard samples available an additional 0.5mL blood sample and a stool sample will be collected on a monthly basis until the subject is discharged from the hospital or up to a maximum of 6 months.
  If the investigators learn information that might be important for the subject's family the investigators may be able to have these results confirmed by a CLIA-certified clinical laboratory that is allowed to provide results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm Infants: Blood samples will be obtained from preterm and former preterm infants at birth and then monthly until hospital discharge. The sample would consist of either up to 0.5ml of blood obtained during a requested clinical blood draw, discarded blood, or a dried blood spot specimen. If no discard samples are available and study blood samples need to be obtained instead, this will occur for a maximum period of 6 months and no more than 3ml of blood will be collected over the entire study period.
- Term Infants: Blood samples will be obtained from term control infants admitted to the NICU monthly until hospital discharge. The sample would consist of either up to 0.5ml of blood obtained during a requested clinical blood draw, discarded blood, or a dried blood spot specimen. If no discard samples are available and study blood samples need to be obtained instead, this will occur for a maximum period of 6 months and no more than 3ml of blood will be collected over the entire study period.

SUMMARY:
The aims of this study are to:

* Assess whether ex-preterm infants have a persistently immature immune system, which may decrease their ability to respond to infections, when they reach term-corrected gestational age.
* Examine whether clinical history, nutrition status, and microbiome composition are linked to the immune composition of term and ex-preterm infants and whether these variables can be used to predict the risk of developing sepsis or having an immunologic disease.

DETAILED DESCRIPTION:
Preterm infants have increased numbers of viral infections in childhood. They are also more likely to die from infection during the neonatal and infant periods than infants born at term. While studies have demonstrated that premature infants have decreased adaptive and innate immune responses compared with infants born at term, there has been little investigation into whether this impaired immunity improves and becomes similar to full term infants once the ex-preterm infants reach term-corrected gestational age. There have likewise not been studies to determine whether specific immune markers may predict the risk of developing sepsis. Given the immaturity of the preterm immune system and the many potential infectious and inflammatory insults they are exposed to during the preterm period (infections, poor nutrition, stress, steroid therapy), there is also a possibility that the relative immune deficiency experienced by preterm infants may persist into infancy.

The goal of this study is to determine whether former preterm infants have sustained differences in immunity compared to age-matched controls, which would have significant implications for infection risk and response to vaccination. Additionally, this study hopes to examine whether certain immune system abnormalities make certain babies more likely to have a serious infection. The present study will assess composition and function of T and B cell compartments in preterm and former preterm infants.

ELIGIBILITY:
Inclusion Criteria Ex-Preterm Infant Group:

* Infants born less than 37 weeks gestational age

Exclusion Criteria for Ex-Preterm Infant Group:

* Infants born greater than 37 weeks gestational age

Inclusion Criteria for Term Infant Group:

* Infants born greater than 37 weeks gestational age

Exclusion Criteria for Term Infant Group:

* Infants born less than 37 weeks gestational age

Ages: 0 Days to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Both term and preterm infants will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The presence or absence of skewed or altered immune profile in preterm infants compared to infants born at term. | Up to 1 year
  The present study will assess composition and function of T and B cell compartments in preterm and former preterm infants. Whole blood samples will be separated into serum and cellular components and sera will be used to assess cytokine predominance and measure nutritional markers.

SECONDARY OUTCOMES:
Determining whether non-modifiable variables of nutrition status, microbiome composition, or immune repertoire composition predict risk of developing infection during the hospitalization. | Up to 1 year
  The investigators will measure nutritional status. Whole blood samples will be separated into serum and cellular components and sera will be used to assess cytokine predominance and measure nutritional markers.

CONTACTS AND LOCATIONS:
Overall Officials: Amy O'Connell, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No